CLINICAL TRIAL: NCT00347685
Title: Open-label Assessment of the Safety and Effectiveness of Extended Release Tramadol (Tramadol ER) in the Treatment of Chronic Non-malignant Pain.
Brief Title: A One-year, Open-label Study to Assess the Safety and Effectiveness of Extended Release Tramadol HCl in the Treatment of Chronic, Non-malignant Pain.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B00.CTOL.003.TRA P03
Record Dates: First submitted 2006-07-01; First posted 2006-07-04 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Pain
Keywords: chronic non-malignant pain; chronic pain; non-malignant; pain; moderate pain; severe pain
MeSH Terms: conditions — Chronic Pain; Pain

INTERVENTIONS:
Drug: tramadol ER

SUMMARY:
The purpose of this study is to assess the safety of tramadol HCl ER following long-term treatment. The study hypothesis is that long-term treatment with tramadol HCl ER is safe and effective for the treatment of chronic, non-malignant pain.

DETAILED DESCRIPTION:
Immediate release (IR) tramadol has demonstrated efficacy in several pain conditions including: obstetrical, gynecological, orthopedic, abdominal, and oral surgery. The short elimination half-life of IR tramadol necessitates every 4-6 hour dosing to maintain optimum levels of analgesia in chronic pain. The study medication in this study is a once-daily, extended release (ER) tramadol formulation. This study is a multicenter, multiple-dose, 1-year open-label study designed to assess the safety and effectiveness of tramadol HCl ER. Patients with moderate to severe chronic non-malignant pain, requiring treatment with an analgesic on a daily basis, are eligible for study participation. Patients eligible for enrollment are as follows: those who completed 12 weeks in one of two prior double-blind studies ("roll-over patients") or those without participation in any prior study of tramadol HCl ER ("direct enrollment patients"). Following a screening evaluation and baseline assessment, roll-over patients will be treated for up to 38 weeks and direct enrollment patients for up to 58 weeks. At baseline (Visit 2), patients will receive tramadol HCl ER 100 mg once daily (QD) for 3 days; on day 4, they will increase to tramadol HCl ER 200 mg QD, based on tolerability. Patients will be required to be on a minimum dose of tramadol HCl ER 200 mg QD by Visit 3. At Visit 4, patients are required to begin treatment with a minimum dose of tramadol HCl ER 300 mg QD. The maximum dose of tramadol HCl ER for patients >= 75 years old is 300 mg QD. By Visit 5, patients < 75 years old are to be initiated on a tramadol HCl ER dose of 400 mg QD. Patients who cannot tolerate a dose increase of tramadol HCl ER from 300 mg or 400 mg QD (due to side effects) or who upon dose increase cannot tolerate the dose will be permitted to reduce the tramadol HCl ER dose to 300 mg QD. Patients unable to tolerate tramadol HCl ER 300 mg or 400 mg QD or those who had pain unresponsive to appropriate dose adjustments will be discontinued and alternate analgesic therapy initiated, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of chronic, non-malignant pain >= 6 months requiring treatment with an analgesic; females of childbearing potential practicing abstinence or a medically accepted form of contraception with a negative serum pregnancy test within 7 days of study entry; patients able to understand the procedures, complete the pain scales and able to communicate meaningfully with study personnel; patients who agree to study participation and sign a form indicating their informed consent.

Exclusion Criteria:

* Patients with an uncontrolled medical condition; patients whose weight <= 100 pounds; patients with dysphagia or difficulty swallowing tablets; patients with intractable nausea and vomiting; patients with a history of clinically significant intolerance to tramadol or a known hypersensitivity to opioid analgesics, such that treatment with tramadol or other opioids is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650
Dates: Start 2000-10; Study Completion 2003-02

PRIMARY OUTCOMES:
The primary outcomes are analyses of adverse events (incidence, frequency,
severity, attribution, adverse events causing withdrawal from study)

SECONDARY OUTCOMES:
The secondary outcomes are pain intensity (visual analog scale) assessment,
patient global assessment of study medication, pain recall (least, worst and
average pain); changes from baseline to each subsequent visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Gainesville Clinical Research Center, Gainesville, Florida, United States